CLINICAL TRIAL: NCT01303133
Title: Natural History of Amyloid Deposition in Adults With Down Syndrome
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Benjamin L Handen, PhD, BCBA-D, Principal Investigator, University of Pittsburgh
Other Study IDs: PRO09080266; 2R01AG031110-03A1 (NIH); NCT01412255 (obsolete NCT alias)
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Down Syndrome
Keywords: beta amyloid, Down Syndrome, Alzheimer's Disease
MeSH Terms: conditions — Down Syndrome; Plaque, Amyloid; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Trisomy 21 ApoE
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Adults with Down Syndrome ages 30+ (PiB-/-): We will be recruiting healthy adults with Down syndrome ages 30 and over. Participants cannot have a diagnosis of dementia.
- Adults with Down Syndrome ages 30+ (PiB-/+)
- Adults with Down Syndrome ages 30+ (PiB+/+)

SUMMARY:
The primary objective of this study is to assess the presence of amyloid in non-demented/functionally stable adults with DS as a function of age, dividing the sample into amyloid-positive and amyloid-negative groups. We will also obtain baseline cognitive measures across a range of areas that are often affected by AD.

DETAILED DESCRIPTION:
Specific Aim 1: To assess and compare amyloid deposition (with PiB PET) in non-demented/functionally stable adults with DS across three age cohorts (30-39, 40-49, and >50 years of age).

Primary Hypothesis 1: At initial assessment, there will be a significantly higher prevalence of amyloid-positive (PiB+) subjects in each succeeding age cohort.

In addition, we will test the following secondary hypothesis:

Secondary Aim 1: To compare the presence or absence of the apolipoprotein-E4 allele to the retention of PiB in various brain areas of the DS subjects.

Secondary Hypothesis 1: At baseline, subjects who carry at least one Apolipoprotein-E4 (ApoE4) allele will show a higher prevalence of being PiB+.

ELIGIBILITY:
Inclusion Criteria:

1. Participant IQ at least 47 (based upon Stanford-Binet V Abbrev. Test Battery)
2. Participant at least 30 years of age
3. DSDS score indicating participant is asymptomatic for AD
4. Reliable caregiver who is capable of providing correct information about the participant's clinical symptoms and history
5. Agreement of caregiver and clinician that participant is able to cooperate with the protocol tasks
6. Participant has provided assent (or consent) and/or parent/caregiver has provided informed consent

Exclusion Criteria:

1. Participant is non-verbal or has extremely limited language skills
2. Score within the "symptomatic" range on the DSDS
3. Any significant disease or unstable medical condition that could affect neuropsychological testing
4. Any problems with vision or hearing that could affect neuropsychological testing
5. Participants in whom MRI is contraindicated
6. Claustrophobia or prior failed experiences of completing MRI scans or blood draws
7. Participant is pregnant or breast feeding
8. History or other evidence of severe illness or other condition that would make the participant, in the opinion of the investigator, unsuitable for the study?

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non-Demented Adults with Down Syndrome, ages 30 and above
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2009-08; Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Amyloid deposition | every 36 months for 9 years
  Obtained via PiB PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Handen, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh and University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Waisman Center at the University of Wisconsin - Madison, Madison, Wisconsin